CLINICAL TRIAL: NCT07151287
Title: Diagnosis of Intracranial Hypertension Using TCCD, ONSD and ODH by Bedside Ultrasound
Status: Not yet recruiting | Type: Observational
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Jinfang Liu, MD, Director of the Neurotrauma and Neurointensive Care Group, Xiangya Hospital of Central South University
Other Study IDs: Ultrasound-ICP
Record Dates: First submitted 2025-07-02; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury
Keywords: traumatic brain injury; craniocerebral trauma; brain trauma; intracranial pressure; transcranial Doppler ultrasound
MeSH Terms: conditions — Brain Injuries, Traumatic; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with traumatic brain injury and invasive ICP monitoring: Patients with traumatic brain injury and invasive ICP monitoring.
  Interventions: Diagnostic Test: TCCD; Diagnostic Test: ONSD; Diagnostic Test: ODH; Diagnostic Test: Invasive ICP

INTERVENTIONS:
Diagnostic Test: TCCD — Patients receive non-invasive assessments of TCCD using bedside ultrasound.
Diagnostic Test: ONSD — Patients receive non-invasive assessments of ONSD using bedside ultrasound.
Diagnostic Test: ODH — Patients receive non-invasive assessments of ODH using bedside ultrasound.
Diagnostic Test: Invasive ICP — Patients receive invasive assessments of ICP.

SUMMARY:
The goal of this observational study is to investigate several means of measuring intracranial pressure (ICP) non-invasively in patients who had head trauma and received implantation of invasive ICP monitor device. The main questions it aims to answer are:

What are the diagnostic efficacies of Transcranial Color-Coded Doppler Ultrasound (TCCD), Optic Nerve Sheath Diameter (ONSD) and Optic Disc Height (ODH) (the 3 non-invasive way of measuring ICP) compared with invasive ICP monitor? Participants will receive simultaneous non-invasive measurements of TCCD, ONSD and ODH along with during the days of invasive ICP monitoring. The data will be compared among the techniques to study the diagnostic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic brain injury;
* Received invasive ICP monitoring;
* age ≥ 18 years old.

Exclusion Criteria:

* Severe eyeball / eyelid damage prevents transorbital ultrasound examination;
* Allergy to ultrasound coupling agent;
* Pregnant or lactating females.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study selects patients admitted to the neurosurgical intensive care unit of Central South University Xiangya Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 64 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity of TCCD | Day 0 (when invasive ICP probe is implanted) to day 10
  Sensitivity and specificity of diagnosing intracranial hypertension using TCCD
Sensitivity and specificity of ONSD | Day 0 (when invasive ICP probe is implanted) to day 10
  Sensitivity and specificity of diagnosing intracranial hypertension using ONSD
Sensitivity and specificity of ODH | Day 0 (when invasive ICP probe is implanted) to day 10
  Sensitivity and specificity of diagnosing intracranial hypertension using ODH

SECONDARY OUTCOMES:
Pearson correlation coefficient between ultrasound metrics and invasive ICP | Day 0 (when invasive ICP probe is implanted) to day 10
  Pearson correlation coefficient between metrics from bedside ultrasound and invasive ICP

IPD SHARING:
Plan to Share IPD: No
Data cannot be shared publicly because of patient privacy protection. Data are available from the Xiangya Hospital Institutional Data Access / Ethics Committee for researchers who meet the criteria for access to confidential data.